CLINICAL TRIAL: NCT00321360
Title: Reaction Time Monitored Patient Maintained Propofol Sedation: a Volunteer Safety Study
Brief Title: Effect Site Controlled, Reaction Time Safeguarded, Patient Maintained Sedation With Propofol in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sonia Allam (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor-Investigator, Sonia Allam, Research Fellow in Anaesthesia, University of Glasgow
Organization: University of Glasgow (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9813
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: propofol; sedation
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Propofol
Device: Patient maintained sedation

SUMMARY:
Whether patient-maintained sedation (the patient controls his/her degree of sedation using a hand-held device) using the drug propofol is safer and more effective when using deteriorating reaction time as an added safeguard against the small potential for over sedation in a group of healthy volunteers.

DETAILED DESCRIPTION:
Patients receiving conscious sedation for dentistry and endoscopy are usually treated with intermittent bolus doses of intravenous midazolam (administered by the operator-sedationist). The safety of such a regime has been questioned with reports of up to 13 % of patients desaturating to below 80 % in the recovery area following sedation for endoscopy. Mortality occurs in 0.05 % of endoscopy patients (with approximately 60 % of this being due to hypoxaemia). The aim of our work, therefore, is to look at providing sedation that is both safer as well as being efficacious.

The drug propofol, the agent most commonly used to induce general anaesthesia in the UK, is also frequently administered intravenously by anaesthetists in low doses to provide conscious sedation for patients undergoing unpleasant procedures i.e. patients become relaxed, anxiety-free, but maintain verbal contact throughout.

The technique of patient maintained sedation using the drug propofol (the patient can increase the amount of sedation (and propofol) they receive by pressing a demand button attached to a standard infusion device) has been used by anaesthetists and evaluated since 1997.

Several recent studies published and submitted for publication by this research group on patient maintained sedation using the drug propofol have shown this method of sedation to be safe and effective in dental patients (over 120 patients studied and no cases of over sedation). It was also shown that this method, when compared to the established method of sedation in oral surgery (the dentist administering doses of midazolam intravenously), produced both quicker recovery and less anxiety prior to the surgery.

The routine use of propofol traditionally is restricted to anaesthetists, as in much higher doses general anaesthesia is produced with possible loss of airway patency. Currently the safety feature is predominantly that as patients become more sedated they cannot press the patient demand button and hence cannot increase the amount of propofol they are receiving. Also the device ensures that the blood and brain concentrations have equilibrated to within 10% of each other before another successful demand for propofol can be made (usually takes approximately two minutes) and it only allows a maximum calculated brain concentration of 3 micrograms/milliliter of propofol. The device also will start to decrease the calculated brain concentration of propofol if the demand button has not been pressed for six minutes.

Despite the encouraging results above we also found in a recent pilot study involving 20 healthy volunteers who were instructed to try and make themselves unconscious that there were 2 cases of over sedation (of these one briefly lost verbal contact and the other required supplemental oxygen for a short time only). This however was not unsafe in the presence of an anaesthetist. Over sedation, however, was never demonstrated with any of the oral surgery patients in the previous studies. This may have been due to a higher level of anxiety in dental patients affecting response to propofol.

We have therefore incorporated an additional safety feature into the existing and previously studied patient maintained sedation system which may further decrease or eliminate this small risk of over sedation. All the above safety features are retained and in addition the patient demand button will now also be used to monitor reaction time at one minutely intervals.

It is known that propofol slows the reaction time of a given individual and in another recent study of 40 patients undergoing general anaesthesia for planned surgery using propofol, the patients' reaction times were recorded both awake and during induction of anaesthesia by instructing the patients to press a handheld button as quickly as possible in response to the handset vibrating. The calculated effect site (brain) concentration of propofol was increased incrementally and reaction time monitored at each stage until the patient could no longer press the button.

The data from this study (deteriorating patient reaction time with increased brain concentration of propofol) was analysed and this information used to provide an additional safeguard within the system to prevent over sedation i.e. a patient's reaction time deterioration by a certain percentage will prevent himself or herself being able to self-administer more propofol. Furthermore the system will actually start to decrease the brain concentration of propofol once the patients' reaction time becomes too slow. The patient demand button will be used to monitor reaction time at one minutely intervals as well as administer more propofol.

We hope that this will eliminate the small risk of over sedation and wish to recruit a further 20 healthy volunteers to assess the safety and efficacy of this reaction time safeguarded, patient-maintained sedation system.

After expressing an interest to be recruited each volunteer will be given the volunteer information leaflet about the research to take home and read. The volunteer will be given ample opportunity to ask any questions regarding the research and to give informed written consent at the study visit.

The volunteer will then have an intravenous cannula sited and will have routine monitoring applied for continuous observation (blood pressure, ECG and oxygen saturation). The cannula will be connected to an effect-site controlled infusion system consisting of a Graseby 3400 infusion pump and a backbar microprocessor (into which the patient's age and weight are entered), programmed with the pharmacokinetic data describing the distribution and elimination of propofol. The microprocessor will also be connected to the investigator's laptop. Whilst the volunteer is connected to the propofol infusion, an experienced anaesthetist (with FRCA qualification) and a trained assistant will be in constant attendance. There will be ready access to all appropriate resuscitation equipment and drugs. Recordings of the patient's vital signs on a data collection sheet will be made prior to sedation and then every 5 minutes until the sedation period ends (see supplements). The anaesthetist will also record the volunteer's sedation score at each reaction time challenge (see supplements). For each reaction time challenge the actual reaction time and corresponding effect site (brain) concentration will be logged onto the laptop.

The way the device works will be explained and the volunteer will be given a handset to hold which has a button on top. They will hold this throughout the procedure. The handset will vibrate at intervals of one minute throughout the procedure and the volunteer will be instructed to press the button twice (double click) as soon as the handset vibrates in order to record the volunteer's reaction time. Three baseline reaction times will be recorded prior to sedation, the first value discarded and the second two values averaged to give the baseline reaction time. We will also tell them that the way to demand more propofol during the sedation period is by also pressing the button twice within one second.

The device will then be set to achieve an effect-site (brain) concentration of 1.0 micrograms/millilitre (mcg/ml). Once this effect concentration has been achieved the control button will be activated for administration of propofol and the volunteer will be instructed to "try to make yourself unconscious". The volunteer can increase the effect site concentration by 0.2 mcg/ml with each successful double press (up to a maximum of 3 mcg/ml).

A double press will only be successful once between reaction time measurements and provided blood and brain concentrations of propofol have equilibrated to within 10% of each other and provided reaction time does not become more prolonged than 150% of the baseline value. In this case no further drug increments will be permitted and effect site concentration will be maintained at the same level for two minutes after which time a successful demand press would only occur if reaction time became less than 150% again. In addition an even more prolonged reaction time of greater than 200% from baseline would actually lead to a reduction in effect site concentration of propofol.

If the volunteer becomes unresponsive to verbal command or reaches the set maximum effect site concentration of 3 mcg/ml, or in the unlikely event the volunteer desaturates to a level below 90% or shows any other signs of respiratory depression, the infusion will be ended. The volunteer will be looked after by the anaesthetist (ensuring that the airway is maintained, supplemental oxygen is given and ventilation is adequate) until awake and responsive to speech and at this point they will be taken to the sedation suite recovery room.

Otherwise the sedation period will end after a 30 minute period or once the device has decreased the brain concentration of propofol on three successive occasions (due to reaction time slowing).

The volunteer will then be transferred to a recovery area, where they will be monitored until ready for discharge according to sedation suite criteria. Just prior to discharge volunteers will complete a short questionnaire to assess recall and satisfaction (see supplements).

As stated on volunteer information leaflet, volunteers can withdraw from the study at any time without giving a reason and without their care being in any way affected.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II (healthy or mild systemic illness) healthy volunteers
* Age 18 - 50

Exclusion Criteria:

* ASA III or above
* Out with age group above
* Contraindication to propofol
* History of epilepsy
* History of substance abuse
* Major Psychiatric illness
* Pregnancy or breastfeeding
* Unable or unwilling to give informed consent
* Unable to use necessary apparatus
* Vulnerable groups

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-05; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Minimal Sedation Level obtained (modified Objective Observer's Assessment of Sedation)
Maximal change in oxygen saturation (SpO2)

SECONDARY OUTCOMES:
The maximal effect site concentration of propofol at which the minimal sedation level and maximal change in oxygen saturation were achieved
Relationship between reaction time, sedation level and effect site concentration of propofol
Requirement for supplementary oxygen (if SpO2 < 90%)
Requirement for airway or ventilatory support
Maximal change in heart rate (HR), respiratory rate (RR) and blood pressure (BP)
Volunteer satisfaction and recollection

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Allam, MB ChB FRCA, Principal Investigator — University of Glasgow Dept of Anaesthesia
Locations (1):
- Glasgow Dental Hospital, Glasgow, Strathclyde, United Kingdom